CLINICAL TRIAL: NCT04060862
Title: A Phase Ib/III Study of Ipatasertib Plus Palbociclib and Fulvestrant Versus Placebo Plus Palbociclib and Fulvestrant in Hormone Receptor Positive and HER2 Negative Locally Advanced Unresectable or Metastatic Breast Cancer
Brief Title: A Study of Ipatasertib Plus Palbociclib and Fulvestrant Versus Placebo Plus Palbociclib and Fulvestrant in Hormone Receptor Positive and HER2 Negative Locally Advanced Unresectable or Metastatic Breast Cancer
Acronym: IPATunity150
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to not open the Phase III portion was based on a strategic sponsor decision and not driven by any safety concerns.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO41012; 2019-001072-11 (EudraCT Number)
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; palbociclib; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b and Phase 3: Ipatasertib + Palbociclib +Fulvestrant (Experimental)
  Interventions: Drug: Ipatasertib; Drug: Palbociclib; Drug: Fulvestrant
- Phase 3: Placebo + Palbociclib + Fulvestrant (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Ipatasertib — Phase 1b: Ipatasertib, 300 mg starting dose administered orally once daily (PO QD) during an initial 5-7 day run-in period, then continued on Days 1-21 during the first cycle. Starting with Cycle 2, Day 1 ipatasertib will be taken orally once daily on Days 1-21 of each 28-day cycle. Phase 3: Ipatasertib, administered PO QD on Days 1-21 of each 28-day cycle at the dose confirmed in the Phase Ib portion.
  Other Names: RO5532961, GDC-0068
  Arms: Phase 1b and Phase 3: Ipatasertib + Palbociclib +Fulvestrant
Drug: Placebo — Phase 3: Matching placebo, administered PO QD on Days 1-21 of each 28-day cycle at the dose confirmed in the Phase Ib portion.
  Arms: Phase 3: Placebo + Palbociclib + Fulvestrant
Drug: Palbociclib — Palbociclib, administered PO QD on Days 1-21 of each 28-day cycle.
Drug: Fulvestrant — Fulvestrant, 500 mg administered as two intramuscular injections of 250 mg each on Cycle 1 Days 1 and 15 and Day 1 of each subsequent 28-day cycle.

SUMMARY:
The open-label Phase Ib portion of this study will evaluate the safety and pharmacokinetics of ipatasertib in combination with palbociclib and fulvestrant to identify a dose of ipatasertib that can be combined with palbociclib and fulvestrant in the Phase III portion. The randomized Phase III portion of this study will evaluate the efficacy, safety, and patient-reported outcome (PRO) objectives of ipatasertib + palbociclib + fulvestrant compared with placebo + palbociclib + fulvestrant in patients with HR+ HER2-, locally advanced unresectable or metastatic breast cancer who had relapsed during adjuvant endocrine therapy or progressed during the initial 12 months of first-line endocrine therapy in locally advanced unresectable or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* HR+ HER2- adenocarcinoma of the breast that is locally advanced unresectable or metastatic
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating sperm
* Radiologic/objective relapse during adjuvant endocrine therapy or disease progression during the initial 12 months of 1L endocrine therapy in locally advanced unresectable or metastatic breast cancer
* At least one measurable lesion via Response Evaluation Criteria in Solid Tumors, Version 1.1
* Phase III only: Tumor specimen from the most recently collected, available tumor tissue

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant
* Prior treatment with fulvestrant or other selective estrogen receptor down-regulator
* Prior treatment with PI3K inhibitor, mTOR inhibitor or AKT inhibitor
* Phase III only: Prior treatment with CDK4/6 inhibitor for locally advanced unresectable or metastatic breast cancer
* Prior treatment with a cytotoxic chemotherapy regimen for metastatic breast cancer
* History of Type I or Type II diabetes mellitus requiring insulin
* History of or active inflammatory bowel disease or active bowel inflammation
* Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (5):
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute; GYN Oncology, Boston, Massachusetts
  - Summit Medical Group; MD Anderson Cancer Center, Florham Park, New Jersey
- Australia (2):
  - Cabrini Medical Centre; Oncology, Malvern, Victoria
  - Sunshine Hospital, St Albans, Victoria
- Brazil (2):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
- Canada (3):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Juravinski Cancer Clinic; Clinical Trials Department, Hamilton, Ontario
  - Hopital du Saint Sacrement, Québec, Quebec
- Japan (2):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kanagawa Cancer Center, Kanagawa
- Asan Medical Center, Seoul, South Korea
- Spain (2):
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
- United Kingdom (3):
  - The Royal Marsden Hospital; Dept of Medicine, London
  - Christie Hospital NHS Trust, Manchester
  - Royal Marsden Hosp NHS Fnd; Medicine - Breast Unit, Sutton

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study at 12 investigative centers in 7 countries from 21 November 2019 to 29 August 2023.
Pre-assignment Details: This study was planned to include two phases - Phase Ib and Phase III. No participant was enrolled in Phase III as the study was terminated early.
Groups:
- Phase Ib: Ipatasertib + Palbociclib +Fulvestrant: Participants received ipatasertib 300 mg orally (PO) once daily (QD) during an initial 5-7 day during run-in and thereafter on Days 1-21 of each cycle (Cycle length= 28 days) along with palbociclib, 125 mg PO QD on Days 1-21 of each cycle and fulvestrant, 500 mg, intramuscularly (IM) on Days 1 and 15 of Cycle 1 and then on Day 1 of each subsequent cycle for a maximum of 35 months. Only the first 10 participants received single agent ipatasertib during the initial 5-7 day safety run-in. After safety assessment of the run-in participants, further participants were enrolled in this arm to start receiving study treatments on Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant
Started | 20
Completed | 0
Not Completed | 20
Not completed — Symptomatic Deterioration | 1
Not completed — Un-specified | 6
Not completed — Progressive disease | 12
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all the enrolled participants.
Groups:
- Phase Ib: Ipatasertib + Palbociclib +Fulvestrant: Participants received ipatasertib 300 mg PO QD during an initial 5-7 day run-in, and thereafter on Days 1-21 of each cycle (Cycle length= 28 days) along with palbociclib, 125 mg PO QD on Days 1-21 of each cycle and fulvestrant, 500 mg, IM on Days 1 and 15 of Cycle 1 and then on Day 1 of each subsequent cycle for a maximum of 35 months. Only the first 10 participants received single agent ipatasertib during the initial 5-7 day safety run-in. After safety assessment of the run-in participants, further participants were enrolled in this arm to start receiving study treatments on Cycle 1 Day 1.
Arm/Group | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase III: Progression-Free Survival (PFS), as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurred first. Progressive disease (PD) is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of ≥ 5 millimeters (mm).
Time Frame: From randomization in Phase III until the first occurrence of disease progression or death from any cause, whichever occurs first, up to approximately 36 months
Population: The study was terminated before initiation of Phase III as per sponsor's decision; hence this outcome measure was not assessed or analyzed, and no data collected.
Groups:
- Phase III: Ipatasertib + Palbociclib +Fulvestrant: Ipatasertib, 300 mg PO QD along with palbociclib, 125 mg PO QD on Days 1-21 of each 28-day cycle and fulvestrant, 500 mg, IM injections on Days 1 and 15 of Cycle 1, then on Day 1 of each subsequent 28-day cycle until progressive disease (PD) or unacceptable toxicity, whichever occurs first.
- Phase III: Placebo + Palbociclib + Fulvestrant: Placebo PO QD along with palbociclib, 125 mg PO QD on Days 1-21 of each 28-day cycle and fulvestrant, 500 mg IM injection on Days 1 and 15 of Cycle 1, then on Day 1 of each subsequent 28-day cycle until PD or unacceptable toxicity, whichever occurs first.
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Phase Ib: Number of Participants With Adverse Events and Adverse Events With Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: AE=any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. Severity of AEs were rated per NCI CTCAE v5 where, Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental Activities of Daily Living (ADL); Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL; Grade 4 Life-threatening consequences; urgent intervention indicated; Grade 5 Death related to AE.
Time Frame: Up to 36 Months
Population: Safety evaluable population included all randomized participants who received any amount of study drug (i.e., ipatasertib + palbociclib + fulvestrant).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Ipatasertib + Palbociclib +Fulvestrant: Participants received ipatasertib 300 mg PO QD during an initial 5-7 day run-in, and thereafter on Days 1-21 of each cycle (Cycle length= 28 days) along with palbociclib, 125 mg PO QD on Days 1-21 of each cycle and fulvestrant, 500 mg, IM on Days 1 and 15 of Cycle 1 and then on Day 1 of each subsequent cycle for a maximum of 35 months. Only the first 10 participants received single agent ipatasertib during the initial 5-7 day safety run-in. After safety assessment of the run-in participants, further participants were enrolled in this arm to start receiving study treatments on Cycle 1 Day 1.
Arm/Group | Phase 1b: Ipatasertib + Palbociclib +Fulvestrant
Number analyzed (Participants) | 20
Participants
  Any AE: Any Grade | 20
  Grade 1 | 3
  Grade 2 | 3
  Grade 3 | 12
  Grade 4 | 5

3. Secondary Outcome: Phase Ib: Plasma Concentration of Ipatasertib and Its Metabolite G-037720
Description: Plasma concentrations of Ipatasertib and its metabolite G-037720 are reported.
Time Frame: Cycle 1, Day 1 and 15: 0.25 hours pre-dose, 0.5, 1, 2, 3, 4 and 6 hours post- dose ; Cycle 2, Day 15: 0.25 hours pre-dose; Cycle 3, Day 15: 0.15 hours pre-dose, 2 hours post-dose (each cycle = 28 days)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received study treatment. Number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1b: Ipatasertib + Palbociclib +Fulvestrant
Number analyzed (Participants) | 20
nanograms per milliliter (ng/mL)
  Ipatasertib: Cycle 1 Day 15 0.25 hours pre-dose | 46.6 (56.0)
  Ipatasertib: Cycle 1 Day 15 0.5-hours post-dose | 150 (112.3)
  Ipatasertib: Cycle 1 Day 15 1-hours post-dose | 236 (83.4)
  Ipatasertib: Cycle 1 Day 15 2-hours post-dose | 299 (68.0)
  Ipatasertib: Cycle 1 Day 15 3-hours post-dose: number analyzed (Participants) | 19
  Ipatasertib: Cycle 1 Day 15 3-hours post-dose | 290 (34.2)
  Ipatasertib: Cycle 1 Day 15 4-hours post-dose: number analyzed (Participants) | 19
  Ipatasertib: Cycle 1 Day 15 4-hours post-dose | 244 (30.2)
  Ipatasertib: Cycle 1 Day 15 6-hours post-dose: number analyzed (Participants) | 19
  Ipatasertib: Cycle 1 Day 15 6-hours post-dose | 192 (40.1)
  Ipatasertib: Cycle 2 Day 15 0.25 hours pre-dose: number analyzed (Participants) | 17
  Ipatasertib: Cycle 2 Day 15 0.25 hours pre-dose | 42.8 (46.4)
  Ipatasertib: Cycle 3 Day 15 0.15 hours pre-dose: number analyzed (Participants) | 19
  Ipatasertib: Cycle 3 Day 15 0.15 hours pre-dose | 37.6 (58.3)
  Ipatasertib: Cycle 3 Day 15 2-hours post-dose: number analyzed (Participants) | 18
  Ipatasertib: Cycle 3 Day 15 2-hours post-dose | 258 (40.8)
  G-037720: Cycle 1 Day 15 0.25 hours pre-dose | 22.9 (69.3)
  G-037720: Cycle 1 Day 15 0.5-hours post-dose | 38.2 (82.5)
  G-037720: Cycle 1 Day 15 1-hour post-dose | 74.1 (96.3)
  G-037720: Cycle 1 Day 15 2-hours post-dose | 110 (74.0)
  G-037720: Cycle 1 Day 15 3-hours post-dose: number analyzed (Participants) | 19
  G-037720: Cycle 1 Day 15 3-hours post-dose | 116 (47.6)
  G-037720: Cycle 1 Day 15 4-hours post-dose: number analyzed (Participants) | 19
  G-037720: Cycle 1 Day 15 4-hours post-dose | 99.9 (47.9)
  G-037720: Cycle 1 Day 15 6-hours post-dose: number analyzed (Participants) | 19
  G-037720: Cycle 1 Day 15 6-hours post-dose | 81.2 (52.7)
  G-037720: Cycle 2 Day 15 0.25 hours pre-dose: number analyzed (Participants) | 17
  G-037720: Cycle 2 Day 15 0.25 hours pre-dose | 17.5 (45.6)
  G-037720: Cycle 3 Day 15 0.15 hours pre-dose: number analyzed (Participants) | 19
  G-037720: Cycle 3 Day 15 0.15 hours pre-dose | 16.4 (45.2)
  G-037720: Cycle 3 Day 15 2-hours post-dose: number analyzed (Participants) | 18
  G-037720: Cycle 3 Day 15 2-hours post-dose | 92.5 (40.1)

4. Secondary Outcome: Phase Ib: Maximum Concentration (Cmax) of Ipatasertib and Its Metabolite G-037720 in Plasma
Description: Cmax of ipatasertib and its metabolite G-037720 in plasma is reported.
Time Frame: Cycle 1: Day 1 and Day 15
Population: PK-evaluable population included all participants who received study treatment. Overall number analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant
Number analyzed (Participants) | 9
ng/mL
  Ipatasertib: Cycle 1 Day 1 | 294 (52.6)
  Ipatasertib: Cycle 1 Day 15 | 437 (41.1)
  G-037720: Cycle 1 Day 1 | 120 (84.2)
  G-037720: Cycle 1 Day 15 | 137 (53.4)

5. Secondary Outcome: Phase Ib: Area Under the Plasma Concentration Time-curve From Zero to 24 Hours (AUC0-24) of Ipatasertib and Its Metabolite G-037720
Description: AUC0-24 of Ipatasertib and its metabolite G-037720 is reported
Time Frame: Cycle 1: Day 1 and Day 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms/milliliter (h*ng/mL)
Arm/Group | Phase 1b: Ipatasertib + Palbociclib +Fulvestrant
Number analyzed (Participants) | 9
hour*nanograms/milliliter (h*ng/mL)
  Ipatasertb: Cycle 1 Day 1 | 2169.88 (46.3)
  Ipatasertb: Cycle 1 Day 15 | 3636.97 (33.7)
  G-037720: Cycle 1 Day 1 | 1157.02 (76.6)
  G-037720: Cycle 1 Day 15 | 1391.60 (44.9)

6. Secondary Outcome: Phase Ib: Time to Maximum Concentration (Tmax) of Ipatasertib and Its Metabolite G-037720
Description: Tmax of ipatasertib and its metabolite G-037720 isreported.
Time Frame: Cycle 1: Day 1 and Day 15
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant
Number analyzed (Participants) | 9
hours
  Ipatasertib: Cycle 1 Day 1 | 1.00 [0.50 to 4.00]
  Ipatasertib: Cycle 1 Day 15 | 1.92 [0.50 to 4.00]
  G-037720: Cycle 1 Day 1 | 2.00 [0.97 to 4.00]
  G-037720: Cycle 1 Day 15 | 2.00 [1.00 to 3.08]

7. Secondary Outcome: Phase III: Objective Response Rate (ORR) as Determined by the Investigator According to RECIST v1.1
Description: ORR was defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions ≥4 weeks apart, as determined by the investigator according to RECIST v1.1. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in the short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: From randomization in Phase III up to approximately 36 months
Population: as for outcome 1
Groups:
- Phase III: Ipatasertib + Palbociclib +Fulvestrant: Ipatasertib, 300 mg PO QD along with palbociclib, 125 mg PO QD on Days 1-21 of each 28-day cycle and fulvestrant, 500 mg, IM injections on Days 1 and 15 of Cycle 1, then on Day 1 of each subsequent 28-day cycle until PD or unacceptable toxicity, whichever occurs first.
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase III: Duration of Objective Response (DOR) as Determined by the Investigator According to RECIST v1.1
Description: DOR was defined as time from first occurrence of a documented objective response to the first occurrence of disease progression as determined by investigator per RECIST v1.1, or death from any cause, whichever occurs first. Objective response was defined using RECIST v1.1 criteria as: CR = disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR = at least a 30% decrease in sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in absence of CR. PD = at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to relative increase of 20%, sum of diameters must also demonstrate an absolute increase of ≥ 5 mm. Stable disease (SD): Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase III: Clinical Benefit Rate (CBR) as Determined by the Investigator According to RECIST v1.1
Description: CBR was defined as the percentage of participants who had a CR or PR, or SD for at least 24 weeks, as determined by the investigator according to RECIST v1.1. CR is defined as disappearance of all target lesions. Any pathological lymph nodes must have a reduction in the short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD is defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD is at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of ≥ 5 mm.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase III: Overall Survival (OS) as Determined by the Investigator According to RECIST v1.1
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase III: Time to Deterioration (TTD) in Severity of Pain, According to the Brief Pain Inventory-Short Form (BPI-SF)
Description: TTD in severity of pain is defined as the time from randomization to the first documentation of a 2-point or more increase from baseline on the "worst pain" item from the BPI-SF. A 2-point change is defined as clinically meaningful. The BPI-SF is a widely used patient-reported outcome (PRO) for assessing pain, and the "worst pain" item, frequently used for evaluating increases in the severity of pain. The BPI-SF asks participants to rate their pain at its worst in the last week on a scale from 0 (No pain) to 10 (pain as bad as one can imagine). Higher score indicates more pain.
Time Frame: From randomization in Phase III to the first documentation of a ≥2-point increase in pain scale (up to approximately 36 months)
Population: as for outcome 1
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase III: TTD in Presence and Interference of Pain According to the European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ-C30) Pain Scale
Description: TTD in presence & interference of pain is defined as time from randomization to the first documentation of ≥10-point increase from baseline in EORTC QLQ-C30 pain scale (items 9 & 19). EORTC QLQ-C30 is a validated 30-item self-report measure assessing 5 aspects of participant functioning (physical, emotional, role, cognitive, & social), eight symptom scales (fatigue, nausea & vomiting, pain, dyspnea, insomnia, appetite loss, constipation, & diarrhea), financial difficulties, & global health status/quality of life (GHS/QoL) with a recall period of the previous week. Functioning & symptoms items are scored on a 4-point scale (1=Not at All to 4=Very Much). Pain scale is scored on a 4-point scale (1=Not at All to 4=Very Much) including Item 9: have you had pain? and Item 19: did pain interfere with your daily activity? both range from 1=Not at All to 4=Very Much. All sub-scores are linearly transformed to a total score range of 0-100. Higher scores indicate worse pain symptoms.
Time Frame: From randomization in Phase III to the first documentation of a ≥10-point increase (up to approximately 36 months)
Population: as for outcome 1
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase III: TTD in Physical Functioning (PF), Role Functioning (RF), GHS/QoL According to EORTC QLQ-C30
Description: TTD in PF, RF and GHS/QoL is defined as the time to first documented ≥10-point decrease from baseline in following scales of the EORTC QLQ-C30: PF, RF and GHS/QoL. EORTC QLQ-C30 is a validated 30-item self-report measure assessing 5 aspects of participant functioning (physical, emotional, role, cognitive, & social), eight symptom scales (fatigue, nausea & vomiting, pain, dyspnea, insomnia, appetite loss, constipation, & diarrhea), financial difficulties, & GHS/QoL with a recall period of the previous week. The PF scale has 5 questions about participants' physical functioning and is scored on a 4-point scale (1=Not at All to 4=Very Much). The RF scale is scored on a 4-point scale (1=Not at All to 4=Very Much). The GHS/QoL scale has 7 possible scores of responses (1=Very Poor to 7=Excellent). All sub-scores are linearly transformed to a total score range of 0-100. Higher scores indicate a higher response level (better functioning/QoL).
Time Frame: From randomization in Phase III to the first documentation of a ≥10-point decrease in the PF, RF and GHS/QoL of EORTC QLQ-C30 (up to approximately 36 months)
Population: as for outcome 1
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Phase III: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product; any new disease or exacerbation of an existing disease; recurrence of an intermittent medical condition; any deterioration in a laboratory value or other clinical test; AEs that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment.
Time Frame: Up to approximately 36 months
Population: No data was collected because the study was terminated before the initiation of Phase III per the sponsor's decision.
Arm/Group | Phase III: Ipatasertib + Palbociclib +Fulvestrant | Phase III: Placebo + Palbociclib + Fulvestrant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: Safety evaluable population included all randomized participants who received any amount of study drug (i.e., ipatasertib + palbociclib + fulvestrant).
Arm/Group | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant (N=20)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib: Ipatasertib + Palbociclib +Fulvestrant (N=20)
Anaemia (Blood and lymphatic system disorders) | 8 (13)
Neutropenia (Blood and lymphatic system disorders) | 9 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 17 (70)
Dyspepsia (Gastrointestinal disorders) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (25)
Stomatitis (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 10 (13)
Application site pain (General disorders) | 1 (1)
Asthenia (General disorders) | 8 (8)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Influenza like illness (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (2)
Influenza (Infections and infestations) | 1 (1)
Injection site infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Varicella zoster virus infection (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (6)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (3)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 8 (20)
Platelet count decreased (Investigations) | 6 (22)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (10)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Paresis (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulite (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 8 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 1 (2)
Thrombosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated before initiation of Phase III as per sponsor's decision; hence no primary efficacy and secondary efficacy, safety and pharmacokinetic outcome measures were assessed or analyzed, and no data was collected for Phase III.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT04060862/Prot_SAP_000.pdf